CLINICAL TRIAL: NCT06825494
Title: An Open-label Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of LM-108 ± Penpulimab + Chemotherapy in Patients With Advanced Solid Tumors - Cohort A
Brief Title: Clinical Studies for the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LM-108-Ib/II-01-A
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LM-108 injection+Penpulimab+ Oxaliplatin+Capecitabine (Experimental): LM-108 injection: Intravenous infusion, administered once on Day 1 of each treatment cycle, 21 days as a treatment cycle.
  Penpulimab: Intravenous infusion, administered once on day 1 of each treatment cycle, 21 days as a treatment cycle.
  Oxaliplatin: intravenous infusion over 2 hours once on day 1 of each treatment cycle, 21 days as a treatment cycle.
  Capecitabine: Swallow with water within 30 minutes of meals. Dosing from day 1 to day 14, 2 times a day (1 time in the morning and 1 time in the evening; equal to the total daily dose of 2000 mg/m2); or 1 dose in the afternoon on day 1, 2 times a day from day 2 to day 14, and 1 dose in the morning on day 15. 21 days as a treatment cycle.
  Tislelizumab+Oxaliplatin+Capecitabine
  Interventions: Drug: LM-108 injection+Penpulimab+ Oxaliplatin+Capecitabine
- Tislelizumab+Oxaliplatin+Capecitabine (Experimental): Tislelizumab: intravenous infusion once on day 1 of each treatment cycle,21 days as a treatment cycle.
  Oxaliplatin: intravenous infusion over 2 hours once on day 1 of each treatment cycle, 21 days as a treatment cycle.
  Capecitabine: Swallow with water within 30 minutes of meals. Dosing from day 1 to day 14, 2 times a day (1 time in the morning and 1 time in the evening; equal to the total daily dose of 2000 mg/m2); or 1 dose in the afternoon on day 1, 2 times a day from day 2 to day 14, and 1 dose in the morning on day 15. 21 days as a treatment cycle.
  Interventions: Drug: Tislelizumab+Oxaliplatin+Capecitabine
- LM-108 injection 10mg/kg +penpulimab (Experimental): LM-108injection : Intravenous infusion, administered once on Day 1 of each treatment cycle, once every 3 weeks.
  Penpulimab:Intravenous infusion,administered once on day 1 of each treatment cycle, once every 3 weeks.
  Interventions: Drug: LM-108 injection 10mg/kg +penpulimab
- LM-108 injection 600mg + penpulimab (Experimental): LM-108injection : Intravenous infusion, administered once on Day 1 of each treatment cycle, 21 days as a treatment cycle.
  Penpulimab:Intravenous infusion,administered once on day 1 of each treatment cycle, 21 days as a treatment cycle.
  Interventions: Drug: LM-108 injection 600mg + penpulimab
- Penpulimab+ Oxaliplatin+Capecitabine (Experimental): Penpulimab: Intravenous infusion, administered once on day 1 of each treatment cycle, 21 days as a treatment cycle.
  Oxaliplatin: intravenous infusion over 2 hours once on day 1 of each treatment cycle, 21 days as a treatment cycle.
  Capecitabine: Swallow with water within 30 minutes of meals. Dosing from day 1 to day 14, 2 times a day (1 time in the morning and 1 time in the evening; equal to the total daily dose of 2000 mg/m2); or 1 dose in the afternoon on day 1, 2 times a day from day 2 to day 14, and 1 dose in the morning on day 15. 21 days as a treatment cycle.
  Interventions: Drug: enpulimab+ Oxaliplatin+Capecitabine

INTERVENTIONS:
Drug: LM-108 injection+Penpulimab+ Oxaliplatin+Capecitabine — LM-108 injection is a monoclonal antibody that selectively clears regulatory T cells that infiltrate tumor sites.
  Penpulimab is a novel and differentiated programmed cell death protein 1 (PD-1) monoclonal antibody.
  Oxaliplatin is a third-generation platinum drug. Capecitabine is a fluoropyrimidine.
  Arms: LM-108 injection+Penpulimab+ Oxaliplatin+Capecitabine
Drug: Tislelizumab+Oxaliplatin+Capecitabine — Tislelizumab is a humanized monoclonal antibody against Programmed cell death -Ligand-1(PD-1).
  Oxaliplatin is a third-generation platinum drug. Capecitabine is a fluoropyrimidine.
  Arms: Tislelizumab+Oxaliplatin+Capecitabine
Drug: LM-108 injection 10mg/kg +penpulimab — LM-108injection is a monoclonal antibody that selectively clears regulatory T cells that infiltrate tumor sites.
  Penpulimab is a novel and differentiated programmed cell death protein 1 (PD-1) monoclonal antibody.
  Arms: LM-108 injection 10mg/kg +penpulimab
Drug: LM-108 injection 600mg + penpulimab — LM-108 injection is a monoclonal antibody that selectively clears regulatory T cells that infiltrate tumor sites.
  Penpulimab is a novel and differentiated programmed cell death protein 1 (PD-1) monoclonal antibody.
  Arms: LM-108 injection 600mg + penpulimab
Drug: enpulimab+ Oxaliplatin+Capecitabine — Penpulimab is a novel and differentiated programmed cell death protein 1 (PD-1) monoclonal antibody.
  Oxaliplatin is a third-generation platinum drug. Capecitabine is a fluoropyrimidine.
  Arms: Penpulimab+ Oxaliplatin+Capecitabine

SUMMARY:
This trial is part of a multicenter, open-label Phase Ib/II clinical study evaluating the efficacy, safety, and tolerability of LM-108 in combination with anti-tumor therapy in patients with advanced solid tumors. Phase Ib of Cohort A1 determines the dose of LM-108 in combination with penpulimab + oxaliplatin + capecitabine. Phase II explores the efficacy and safety of LM-108 in combination with anti-tumor therapy in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old.
2. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0-1.
3. At least 1 measurable lesion as determined by RECIST v1.1 assessment. Positron emission tomography (PET) scans and ultrasonography cannot be used for diagnostic purposes.
4. All acute toxicities due to prior antineoplastic therapy or surgery have resolved to Grade 0-1 (according to NCI-CTCAE v5.0) or to the level specified by the enrollment/exclusion criteria. Other toxicities that, in the opinion of the investigator, do not pose a safety risk to the participant, such as alopecia, fatigue, and hearing loss, are excluded.
5. Have adequate organ and bone marrow function, defined below:

   1. Routine blood tests: (no transfusion, no granulocyte colony-stimulating factor (G-CSF), no drug correction) white blood cell count (WBC) ≥ 3,000/mm3 (3.0 × 109/L), neutrophil count (ANC) ≥ 1,500/mm3 (1.5 × 109/L), platelet count (PLT) ≥ 100,000/mm3 (100 × 109/L), hemoglobin (Hb) ≥ 9.0 g/dL (90 g/L);
   2. Biochemical tests: serum albumin ≥ 3.0 g/dL (30 g/L), serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 50 ml/min (calculated using the Cockcroft-Gault formula), total bilirubin (BIL) ≤ 1.5 times the upper limit of normal (ULN); Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) levels ≤ 2.5 times the upper limit of normal (ULN), and patients with liver metastases should ≤ 5× ULN;
   3. The international normalized ratio (INR) is ≤ 1.5, and the prothrombin time (PT) and activated partial thromboplastin time (APTT) are ≤ 1.5 times ULN;
   4. Urine protein< 2+; If the urine protein ≥ 2+, the 24-hour urine protein quantification shows that the protein must be ≤ 1 g;
   5. Cardiac function: left ventricular ejection fraction ≥ 50% on echocardiography.
6. Expected survival ≥ 12 weeks;
7. Non-childbearing is defined as a woman who has reached a postmenopausal state, or who has had a medically documented bilateral oophorectomy. Male participants and female participants of childbearing potential must agree to use 1 medically approved form of contraception for the duration of the trial and for 6 months after the last dose of the trial drug or 9 months after the last dose of the chemotherapy drug (oxaliplatin), whichever is later, and a negative serum pregnancy test within 3 days prior to starting the study drug and not lactating.
8. With the consent of the person and has signed the informed consent form, willing and able to comply with the planned visits, study treatment, laboratory tests, and other trial procedures.

   Enrollment criteria applicable to each cohort:

   Cohorts A1 and A2 must meet the following enrollment criteria:
9. Patients with a pathologically confirmed diagnosis of Gastric cancer (GC) or Gastroesophageal junction cancer (GEJC), evidence of unresectable advanced or metastatic disease, and histologic confirmation of adenocarcinoma.
10. Provide negative reports of human epidermal growth factor receptor 2 (HER2) overexpression or amplification; HER2 overexpression or amplification negative is defined as Immunohistochemistry (IHC) 0/1+, or IHC 2+ with Fluorescence In Situ Hybridization (FISH)/In Situ Hybridization (ISH) negative.
11. No prior systemic therapy (including anti-HER-2 therapy) for advanced or metastatic GC/GEJC. Patients who have received prior adjuvant or neoadjuvant therapy for GC/GEJC (including: chemotherapy, radiotherapy, or chemoradiotherapy) have a time of first recurrence or disease progression greater than 6 months from the end of the last treatment. Participants who have previously received anti-tumor traditional Chinese medicine preparations are allowed, but must be discontinued at least 14 days prior to enrollment.
12. Participants should provide tumor tissue samples: fresh specimens (preferred) or formalin-fixed, paraffin-embedded tumor tissue, or microneedle aspiration tissue collected at radiotherapy-naïve sites within approximately 24 months prior to enrollment (specimens within 6 months prior to the first dose of study drug are recommended and no systemic therapy has been received since the sample was obtained). For participants who are unable to provide tissue samples but meet other enrollment conditions, the investigator and the sponsor will jointly decide whether to enroll.

    Cohorts A3 and A4 need to meet the following enrollment criteria:
13. Patients with pathologically confirmed solid tumors with evidence of advanced or metastatic unresectable disease.
14. Patients with advanced or metastatic solid tumors who have failed at least one prior line of standard therapy. Participants who have previously received anti-tumor traditional Chinese medicine preparations are allowed, but must be discontinued at least 14 days prior to enrollment.

Exclusion Criteria:

1. Microsatellite Instability-High (MSI-H)/deficient Mismatch Repair (dMMR) is known.
2. Presence of uncontrolled or symptomatic active central nervous system metastases that can manifest as the presence of clinical symptoms, cerebral edema, spinal cord compression, carcinomatous meningitis, leptomeningeal disease, and/or progressive growth. Central Nervous System (CNS) metastases may be enrolled in the study if they have been adequately treated (surgical or radiographed) and neurological symptoms have returned to baseline (except for residual signs or symptoms associated with CNS treatment) by at least 14 days prior to enrollment.
3. Pleural effusion and ascites that cannot be controlled after puncture and drainage and other treatments within 14 days prior to enrollment; Pericardial effusion with clinical symptoms or moderate or above.
4. Participant weight loss of more than 20% in 2 months prior to enrollment.
5. Participant weight loss of more than 20% in 2 months prior to enrollment:

   1. Received Chemokine receptor 8 (CCR8) antibody, Cytotoxic T-lymphocyte-Associated Protein-4 (CTLA-4) antibody, or other drugs that act on Treg before enrollment.
   2. Major surgery within 28 days prior to enrollment (tissue biopsy and peripherally venipuncture central venous catheter placement [Peripherally Inserted Central Venous Catheters (PICC)]/port implantation required for diagnosis are permitted).
   3. Use of immunosuppressive medications, excluding nasal spray and inhaled corticosteroids or physiologic doses of systemic steroids (i.e., no more than 10 mg/d prednisone or equivalent pharmacophysiological doses of other corticosteroids) within 14 days prior to enrollment.
   4. Live attenuated vaccine within 28 days prior to enrollment or planned administration during the study and within 60 days after the end of study drug treatment.
   5. Received anti-tumor therapy (including chemotherapy, radiotherapy, immunotherapy, endocrine therapy, targeted therapy, biological therapy, or tumor embolization) within 28 days prior to enrollment.
6. Diagnosis of any other malignancy within 5 years prior to enrollment, except for basal cell carcinoma or squamous cell carcinoma of the skin that can be treated locally and has a clear medical record documented as cured, except for basal cell carcinoma or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, intraductal carcinoma in situ of the breast, and papillary carcinoma of the thyroid gland.
7. Presence of any active, known or suspected autoimmune disease. Participants who are in a stable state and do not require systemic immunosuppressive therapy, such as: type I diabetes mellitus, hypothyroidism requiring only hormone replacement therapy, and skin conditions not requiring systemic therapy (e.g., vitiligo, psoriasis, and alopecia) are allowed.
8. Significant clinically significant bleeding symptoms or definite bleeding tendency within 3 months prior to enrollment; Arterial/venous thrombotic events occurred within 6 months prior to enrollment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism.
9. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to enrollment.
10. Severe, non-healing, or dehiscence wounds and active ulcers or untreated fractures.
11. Presence of grade >1 peripheral neuropathy.
12. Gastrointestinal perforation and/or gastrointestinal fistula within 6 months prior to enrollment;
13. Previous intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction within 6 months prior to enrollment, including incomplete obstruction related to a pre-existing condition or requiring routine parenteral hydration, parenteral nutrition, or tube feeding: Patients may be allowed to be enrolled in the study if at the time of initial diagnosis if the patient has received definitive (surgical) treatment to resolve symptoms.
14. Presence of interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic disease (e.g., diabetes, hypertension, pulmonary fibrosis, acute pneumonia, etc.).
15. Known hypersensitivity to the study drug or any of its excipients; or have had a severe allergic reaction to other monoclonal antibodies.
16. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as Hepatitis B Virus (HBV)-DNA ≥ 500 IU/ml; Hepatitis C, defined as Hepatitis C Virus (HCV)-RNA above the lower limit of detection of the analytical method) or co-infection with hepatitis B and C.
17. Presence of cardiac clinical symptoms or disease that is not well controlled:

    1. Cardiac insufficiency of grade 2 and above according to the New York Heart Association (NYHA) criteria.
    2. Corrected QT Interval (QTc) > 480 ms; The QTc interval was calculated using the Fridericia formula.
    3. Severe/unstable angina.
    4. Myocardial infarction occurred within 12 months prior to enrollment.
    5. Clinically significant supraventricular or ventricular arrhythmias and symptomatic congestive heart failure.
18. Systemic antibiotic use within 28 days prior to enrollment for ≥ 7 days, or unexplained fever >38.5°C during screening/before the first dose (as judged by the investigator, fever due to tumor causes can be enrolled).
19. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
20. Participation in any other drug clinical study within 4 weeks prior to enrollment, or no more than 5 half-lives from the last study drug.
21. Known history of psychotropic substance abuse or drug abuse.
22. Presence of other serious physical or psychiatric illnesses or laboratory abnormalities that may increase the risk of participating in the study, or interfere with the results of the study, and patients who, in the opinion of the investigator, are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events | From first dose to 21days after first dose
  Incidence of Phase Ib DLT events for Cohort A1.
Progression-free survival (PFS) | The estimated time from randomization to patient disease progression was 10 months
  Defined as the time from first dose to first occurrence of disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall response rate (ORR) | The estimated duration was 16 months from enrollment of the first patient to 10 months after enrollment of the last patient
  After enrollment of all patients, the proportion of participants with the best overall efficacy rated as complete response or partial response according to criteria (RECIST1.1).
Duration of response (DOR) | The estimated duration was 16 months from enrollment of the first patient to 10 months after enrollment of the last patient
  Patient from the date of first documentation of objective remission of the tumor to the date of first documentation of objective progression of the tumor or the date of death due to any cause.
Disease control rate (DCR) | The estimated duration was 16 months from enrollment of the first patient to 10 months after enrollment of the last patient
  Proportion of participants with complete response, partial response, and stable disease as rated by RECIST v1.1 criteria for best overall efficacy after enrollment of all patients.
Overall survival (OS) | From randomization until patient death, it is expected to be evaluated up to 5 years
  The time from randomization to death due to any cause.
Number of patients with adverse events (AEs) and serious adverse events (SAEs) | Baseline up to 90 days after the last dose
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
AE/SAE severity | Baseline up to 90 days after the last dose
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Cmax | A1/A2: 0hour in cycle 1, end of LM-108, 4.5hours post penpulimab; 0hour of 2,4,6cycles; 0hour of cycle 9 and every 4cycles. A3/A4: 0hour in cycle 1, end of LM-108, end of penpulimab, 1, 4, 24, 48, 168, 336hour; 0hour of 2, 4, 6cycles. 21 days as a cycle
  The highest blood concentration that occurs after administration.
  A1, A2: cycle1,0 hour, 0 after LM-108, 4.5hours after penpulimab, 0 in 2, 4 and 6 cycles; 0 of cycle9 and every 4 cycles.
  A3, A4: 0hour, instantly after LM-108, and after penpulimab, 1, 4, 24, 48, 168hours, and 336hours after penpulimab, 0 in 2, 4 and 6 cycles. Each cycle is 21 days.
Tmax | A1/A2: 0hour in cycle 1, end of LM-108, 4.5hours post penpulimab; 0hour of 2,4,6cycles; 0hour of cycle 9 and every 4cycles. A3/A4: 0hour in cycle 1, end of LM-108, end of penpulimab, 1, 4, 24, 48, 168, 336hour; 0hour of 2, 4, 6cycles. 21 days as a cycle
  The time it takes to reach the peak concentration after dosing.
T1/2 | A1/A2: 0hour in cycle 1, end of LM-108, 4.5hours post penpulimab; 0hour of 2,4,6cycles; 0hour of cycle 9 and every 4cycles. A3/A4: 0hour in cycle 1, end of LM-108, end of penpulimab, 1, 4, 24, 48, 168, 336hour; 0hour of 2, 4, 6cycles. 21 days as a cycle
  The time it takes for the concentration of the drug to drop by half.
Clearance rate (CL) | A1/A2: 0hour in cycle 1, end of LM-108, 4.5hours post penpulimab; 0hour of 2,4,6cycles; 0hour of cycle 9 and every 4cycles. A3/A4: 0hour in cycle 1, end of LM-108, end of penpulimab, 1, 4, 24, 48, 168, 336hour; 0hour of 2, 4, 6cycles. 21 days as a cycle
  The number of apparent volumes of distribution of the drug cleared from the body per unit of time.
Apparent volume of distribution (Vz) | A1/A2: 0hour in cycle 1, end of LM-108, 4.5hours post penpulimab; 0hour of 2,4,6cycles; 0hour of cycle 9 and every 4cycles. A3/A4: 0hour in cycle 1, end of LM-108, end of penpulimab, 1, 4, 24, 48, 168, 336hour; 0hour of 2, 4, 6cycles. 21 days as a cycle
  The ratio constant of the amount of drug in the body to the concentration of the drug in the blood when the drug reaches homeostasis in the body.
  A1/A2: 0hour in cycle 1, end of LM-108, 4.5hours post penpulimab; 0hour of 2,4,6cycles; 0hour of cycle 9 and every 4cycles. A3/A4: 0hour in cycle 1, end of LM-108, end of penpulimab, 1, 4, 24, 48, 168, 336hour; 0hour of 2, 4, 6cycles. 21 days as a cycle
Incidence of Immunogenicity indicators: anti-drug antibodies (ADA) | 0h on Day 1 of Cycles 1, 2, 4, and 6, 0 hours on Day 1 of Cycle 9 and every 4 cycles thereafter, end of treatment/early withdrawal follow-up, and Safety Follow-up Visit 1 (30 days after last dose). Each cycle is 21 days
  Usually refers specifically to antidrug-binding antibodies.
Incidence of Immunogenicity indicators: neutralizing antibodies (Nab) | 0h on Day 1 of Cycles 1, 2, 4, and 6, 0 hours on Day 1 of Cycle 9 and every 4 cycles thereafter, end of treatment/early withdrawal follow-up, and Safety Follow-up Visit 1 (30 days after last dose). Each cycle is 21 days
  Refers to anti-drug antibodies that interfere with the interaction of a drug with its target.

CONTACTS AND LOCATIONS:
Locations (32):
- China (32):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Peking University Shenzhen Hospita, Shenzhen, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Nanyang Second General Hospital, Nanyang, Henan
  - Ping mei shen ma Medical Group General Hospital, Pingdingshan, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The second xiangya hospital of central south university, Changsha, Hunan
  - Inner Mongolia Hospital of Peking University Cancer Hospita, Hohhot, Inner Mongolia
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - NanJing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - XuZhou Central Hospital, Xuzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital Of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University Medical College, Xi'an, Shaanxi
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shangxi Medical University, Taiyuan, Shangxi
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospita, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Affiliated Cancer Hospital, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang